CLINICAL TRIAL: NCT02375035
Title: Developing a Safer and More Accurate Device for Biopsies of Suspected Prostate Cancer
Acronym: CAMPROBE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Vincent Gnanapragasam, Lecturer in Uro-oncology and Consultant Urological Surgeon, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: AO93224
Record Dates: First submitted 2015-02-19; First posted 2015-03-02 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Prostate Cancer; Prostate Biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: CAMPROBE — To assess patient's experience and complications of the CAMPROBE biopsy needle and compare the results with known published outcomes from standard transrectal biopsies

SUMMARY:
To evaluate the use of the CAMbridge PROstate Biopsy devicE (CAMPROBE) as a method of undertaking prostate biopsy as part of their clinical management.

DETAILED DESCRIPTION:
To assess patient's experience and complications of the CAMPROBE and compare the results with known published outcomes from standard transrectal biopsies .

To use data from the pilot study to determine the feasibility of a randomised trial comparing CAMPROBE with the current standard method of prostate biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Fit and well enough to undergo a repeat prostate biopsy
* Men who have previously had a transrectal ultrasound biopsy of the prostate and due to have a repeat biopsy as part of normal care
* Men on active surveillance
* Men on PSA monitoring

Exclusion Criteria:

* Contraindication for a repeat prostate biopsy
* Contraindication for a transperineal prostate biopsies
* Previous perineal or anal surgery
* MRI suggesting anterior lesion or extra capsular disease
* MRI suggesting lesion that needs fusion image targeting
* Unable to lie down and with legs in a stirrup for at least 45 minutes

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have had a standard biopsy and now require a transrectal biopsy as part of their management
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Pain score assessment of CAMPROBE biopsy procedure | 3 weeks
  Measured using a 10 point visual pain score tool and a point based structured questionnaire
Patient reported adverse events related to CAMPROBE biopsy | 3 weeks
  Point based structured questionnaire assessment of adverse events after biopsy
Patient perception and acceptance of CAMPROBE biopsy | 3 weeks
  Point based structured questionnaire including willingness to recommend to a friend

SECONDARY OUTCOMES:
Deterioration in urinary function after CAMPROBE biopsy | 3 weeks
  Measurement of urinary function after the procedure using a structured questionnaire
Deterioration in sexual function after CAMPROBE biopsy | 3 weeks
  Measurement of urinary function after the procedure using a structured questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Gnanapragasam, Principal Investigator — University of Cambridge
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, United Kingdom